CLINICAL TRIAL: NCT06728865
Title: Evaluation of the Efficacy and Safety of Furmonertinib Combined with Bevacizumab As First-Line Treatment for EGFR-Positive Non-Small Cell Lung Cancer with Brain Metastases: a Single-Arm, Open-Label, Prospective Phase II Clinical Study
Acronym: Better Brain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li-kun Chen (Other)
Responsible Party: Sponsor-Investigator, Li-kun Chen, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10121
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); EGFR Mutation-Positive Lung Cancer; Brain Metastases; Leptomeningeal Metastases; Intracranial Tumor Progression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Meningeal Carcinomatosis | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Furmonertinib Combined with Bevacizumab Treatment Group (Experimental): The treatment regimen is Furmonertinib combined with Bevacizumab.
  Interventions: Drug: The treatment regimen is Furmonertinib combined with Bevacizumab.

INTERVENTIONS:
Drug: The treatment regimen is Furmonertinib combined with Bevacizumab. — The treatment regimen is Furmonertinib combined with Bevacizumab.

SUMMARY:
This study evaluates the safety and efficacy of Befotertinib combined with Bevacizumab as a first-line treatment for patients with EGFR mutation-positive advanced non-small cell lung cancer (NSCLC) accompanied by brain or leptomeningeal metastases. It is a single-arm, open-label, prospective Phase II clinical trial aiming to explore the potential benefits of this combination therapy in improving intracranial progression-free survival (iPFS) and overall survival (OS). Patients will receive Befotertinib daily and Bevacizumab every three weeks until disease progression, intolerable toxicity, or withdrawal of consent. The study seeks to address the unmet need for effective treatments in this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years. ECOG performance status (PS) score of 0-2. Expected survival time of ≥3 months.
2. Histologically or cytologically confirmed non-squamous non-small cell lung cancer (NSCLC).
3. Baseline evaluation confirming the presence of EGFR-sensitizing mutations (19del/L858R) via first- or second-generation sequencing. Test samples can include archived tumor tissue or fresh tumor tissue collected during screening. If unavailable, pleural effusion, cerebrospinal fluid, or blood samples may be used for testing.
4. Asymptomatic brain metastases or those with controlled intracranial hypertension symptoms following dehydration treatment. Continued medication to maintain stable symptoms at enrollment or during the study is allowed.
5. For patients with parenchymal or leptomeningeal brain metastases, MRI must confirm at least one brain lesion with a diameter ≥5 mm.
6. No prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC. Patients who underwent radical surgery, chemoradiotherapy, or adjuvant therapy (chemotherapy or radiotherapy) for early-stage NSCLC may be included if their disease recurred or metastasized after treatment, provided the interval from the last treatment to initial tumor recurrence exceeds 6 months.
7. Normal function of major organs, with the following criteria: Hematology (without transfusion or hematopoietic stimulating factors within 14 days): Hemoglobin (HB) ≥ 90 g/L. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L. Platelets (PLT) ≥ 80 × 10⁹/L. Biochemistry: Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN (if liver metastases are present, ALT and AST < 5 × ULN). Creatinine (Cr) ≤ 1.25 × ULN or creatinine clearance rate (CCr) ≥ 45 mL/min (using the Cockcroft-Gault formula). Proteinuria < 2+ (if baseline proteinuria ≥ 2+, a 24-hour urine protein quantification ≤ 1 g is required). International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN. Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%) as assessed by Doppler ultrasound.
8. Women of childbearing potential must agree to use effective contraception (e.g., intrauterine devices, oral contraceptives, or condoms) during the study and for 6 months after its completion. Negative serum or urine pregnancy test within 7 days prior to enrollment and non-lactating status are required. Male participants must agree to use contraception during the study and for 6 months afterward.
9. Participants must voluntarily consent to participate in the study, sign an informed consent form, and demonstrate good compliance.

Exclusion Criteria:

1. Active Bleeding with Brain and/or Leptomeningeal Metastases
2. Includes therapies with agents such as bevacizumab, endurance, or anlotinib.
3. ≥ Grade 2 toxicity (NCI-CTCAE v4.03) related to prior treatments not resolved at the start of study treatment (excluding alopecia and Grade 2 neurotoxicity caused by platinum agents).
4. Includes uncontrolled nausea/vomiting, inability to swallow, gastrointestinal resection, chronic diarrhea, or intestinal obstruction
5. Prior whole-brain radiotherapy (WBRT). Radiotherapy involving >30% of bone marrow or extensive radiation within 4 weeks before the first dose (palliative radiotherapy for non-brain metastases, such as bone metastases, is exempt).
6. Poorly controlled hypertension (defined as blood pressure ≥160/100 mmHg despite optimal antihypertensive therapy). Cardiac criteria, including: QTcF ≥ 470 msec (average of three ECGs, corrected using Fredericia's formula) at rest. Clinically significant arrhythmias, conduction abnormalities, or ECG changes (e.g., complete left bundle branch block, third-degree AV block, second-degree AV block, PR interval ≥250 msec). Factors increasing risk of QT prolongation or arrhythmias, such as NYHA Class III-IV heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age, or use of QT-prolonging medications. Active or uncontrolled severe infections. Liver disease, including cirrhosis, decompensated liver disease, or chronic active hepatitis. Poorly controlled diabetes (fasting blood glucose >10 mmol/L). Urinalysis showing ≥2+ proteinuria, confirmed by 24-hour urine protein quantification >1.0 g.
7. Presence of unhealed wounds or fractures.
8. NCI-CTCAE > Grade 1 pulmonary bleeding within 4 weeks before enrollment. NCI-CTCAE > Grade 2 bleeding at other sites within 4 weeks before enrollment. Bleeding tendencies (e.g., active gastrointestinal ulcers) or patients on thrombolytic or anticoagulant therapy (e.g., warfarin, heparin, or similar agents).
9. History of arterial/venous thrombosis within 12 months before enrollment, including stroke (e.g., transient ischemic attack, cerebral hemorrhage, or infarction), deep vein thrombosis, or pulmonary embolism.
10. Clinically significant hemoptysis (>50 mL/day) within 3 months before enrollment. Severe bleeding symptoms or conditions such as gastrointestinal bleeding, bleeding gastric ulcers, stool occult blood ≥2+, or vasculitis.
11. History of interstitial lung disease, drug-induced interstitial lung disease, steroid-requiring radiation pneumonitis, or clinically active interstitial lung disease.
12. History of substance abuse or uncontrolled psychiatric disorders.
13. Poorly controlled pleural or ascitic effusions despite symptomatic treatment, causing Grade ≥2 respiratory syndrome (≥CTCAE Grade 2).
14. Known active infections, including: Active hepatitis B (HBsAg positive and HBV-DNA ≥ 2 × 10³ IU/mL during screening). Hepatitis C (HCV-Ab positive and HCV-RNA positive during screening). Active tuberculosis (evidence of active infection within 1 year). Syphilis (both specific and non-specific antibodies positive). HIV infection (HIV antibody positive). Active infections are not routinely screened unless clinically indicated.
15. Severe diseases or conditions deemed to pose risks to patient safety or impede study completion.
16. Severe diseases or conditions deemed to pose risks to patient safety or impede study completion.
17. Prior allogeneic bone marrow transplantation.
18. Prior allogeneic bone marrow transplantation. 19)Any other condition deemed unsuitable for the study by the investigator. 20)Major surgery within 28 days before the first dose (defined as surgeries requiring at least 3 weeks of recovery before study treatment).

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
12-Month Intracranial Progression-Free Survival Rate Assessed by RECIST 1.1 in Patients with EGFR-Mutant NSCLC and Brain Metastases | 12 months from the initiation of treatment
  The primary outcome measure is the 12-month intracranial progression-free survival (iPFS) rate, defined as the proportion of patients who remain free from intracranial disease progression or death due to any cause within 12 months from the initiation of treatment. Disease progression is assessed using the RECIST 1.1 criteria based on imaging studies, including enhanced brain MRI. Progression events are confirmed by independent radiological evaluation to ensure consistency and accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No